



 LSUHSC-NO IRB#: 20-047

Consent Rev. date: 03Apr2020 Protocol Revision #: 31Mar2020, v10

Consent to Participate in a Research Study

KEY INFORMATION FOR: TREATMENT IN PATIENTS WITH SUSPECTED OR CONFIRMED COVID-19 WITH EARLY MODERATE OR SEVERE DISEASE: A RANDOMIZED CLINICAL TRIAL Taking place at: University Medical Center New Orleans, 2000 Canal Street, New Orleans, LA 70112

We are asking you to choose whether or not to participate in a research study about treatment of COVID-19 virus. This page is to give you key information to help you decide whether to participate. We have included detailed information after this page. Please ask the research team any questions you have as you read this document. If you have questions later, the contact information for the research investigator in charge of the study is listed below.

#### WHAT IS THE STUDY ABOUT AND HOW LONG WILL IT LAST?

The purpose of the study is to determine whether the medications used in this study are safe and effective in the treatment of COVID-19. If you agree to participate, you receive one (1) of three (3) possible treatments: hydroxychloroquine (HCQ) OR hydroxychloroquine + azithromycin, OR routine supportive care. Neither HCQ or azithromycin are approved by the FDA for treatment of COVID-19 in the United States. Hydroxycholorquine is an antiviral medication currently approved for the treatment of malaria. Azithromycin is an antibiotic currently approved for the treatment of many bacterial infections.

By doing this study, we hope to learn whether these medications are useful in the treatment of COVID-19 infection. Your participation in this research will last about 30 days.

#### WHAT ARE KEY REASONS YOU MIGHT CHOOSE TO PARTICIPATE IN THIS STUDY?

There is no approved treatment for COVID-19 infection at this time. There is some limited evidence that these medications hold promise in shortening the disease course and decreasing the viral load (amount of virus in a sample of blood). It is possible that there will be no benefit to your participation.

#### WHAT ARE KEY REASONS YOU MIGHT CHOOSE NOT TO PARTICIPATE IN THIS STUDY?

There are risks associated with participation in the study. Common side effects can include:

- Hydroxychloroquine: nausea, vomiting, stomach pain, loss of appetite, weight loss, diarrhea, dizziness, headache, ringing in the ears, mood changes, skin rash, itching, and hair loss
- Azithromycin: diarrhea and nausea

The alternative is not to participate in the study.

#### DO YOU HAVE TO TAKE PART IN THE STUDY?

If you decide to take part in the study, it should be because you really want to participate. You will not lose any services, benefits or rights you would normally have if you choose not to participate.

## WHAT IF YOU HAVE QUESTIONS, SUGGESTIONS OR CONCERNS?

The person in charge of the study is Meredith Clement, MD of the Louisiana State University Health Sciences Center of New Orleans, Department of Infectious Disease. If you have questions, suggestions, or concerns regarding this study or you want to withdraw from the study his/her contact information is: 504-702-3141

If you have questions about your rights as a subject, or want to discuss problems, concerns or questions, or obtain information or offer input, you can contact the Chancellor of the LSU Health Sciences Center of New Orleans at (504) 568-4801.

 LSUHSC-NO IRB#: 20-047

Consent Rev. date: 03Apr2020 Protocol Revision #: 31Mar2020, v10

# LOUISIANA STATE UNIVERSITY HEALTH SCIENCES CENTER in NEW ORLEANS Informed Consent Form

**1. <u>Study Title</u>:** Treatment in Patients with Suspected or Confirmed COVID-19 with Early Moderate or Severe disease: a Randomized Clinical Trial, COVID2020-001

## 2. Performance Sites:

University Medical Center New Orleans, 2000 Canal Street, New Orleans, LA 70112

## 3. Investigators:

Principal Investigator: Meredith Clement, MD

Address: 2000 Canal Street, New Orleans, LA 70112

Phone: 504-702-3141

**24-hour number**: 504-702-3000 (UMCNO operator)

Co-Investigators: Yussef Bennani, MD Jyotsna Fuloria, MD

Address: 2000 Canal Street, New Orleans, LA 70112

Phone: 504-702-3141

In case of a research injury contact: Dr. Clement

Phone: 504-702-3141

#### 4. Purpose of Study:

You have been invited to participate in this research study because you have tested positive for the virus that causes COVID-19. The purpose of the research study is to determine whether use of currently approved antiviral and/or antibiotic medications is safe and effective in the treatment of COVID-19. The study will also determine whether the viral load (amount of virus present in the blood) is decreased with the use of these medications.

The study drugs, hydroxychloroquine and azithromycin, are not FDA approved for the treatment of COVID-19.

## 5. <u>Description of the Study</u>:

This study will take place in the Greater New Orleans area only. About 600 people will take part in this study with LSUHSC-NO and UMCNO.

If you decide to participate in the study, you will be randomized on a 1:1:1 basis to one (1) of three (3) treatments. Randomization means that you have a 1 in 3 chance of receiving any of the treatments listed below.

- Arm A: Control arm routine supportive care
- Arm B: hydroxychloroquine ONLY
  - o Day 1: 400 mg orally twice per day

 LSUHSC-NO IRB#: 20-047

Consent Rev. date: 03Apr2020 Protocol Revision #: 31Mar2020, v10

- $\circ$  Days 2 5: 200 mg orally twice per day
- Arm C: hydroxychloroquine AND azithromycin
  - Day 1: hydroxychloroquine 400 mg orally twice per day AND azithromycin 500 mg orally once per day
  - o Days 2 − 5: hydroxychloroquine − 200 mg orally twice per day AND azithromycin − 250 mg orally once per day

If you decide to participate, this document and the study will be discussed via telephone with you or your legally authorized representative (LAR) before you receive any treatment or have any non-routine care tests performed. This discussion and consent to participation in the study will be documented in your medical record.

<u>Screening/Enrollment/Day1 Tests and Procedures</u> – this visit will occur while you are admitted in the hospital

- Informed consent review
- Randomization to one of the three treatment arms.
- First dose of drug for Arms B and C will be given.
- Your vital signs, height, weight, and medical history will be recorded.
- Blood will be drawn for routine laboratory testing. About 3 tablespoons of blood will be collected.
- Blood or urine will be collected for a pregnancy test if necessary. About 1 tablespoon of blood or 2 tablespoons of urine will be collected.
- An electrocardiogram (ECG) and chest x-ray will be performed if one has not been done up to 1 month before you start the study medication.
- A nasal or oral swab will be taken for testing of the virus.

<u>Day 3, 6, and 14 Tests and Procedures</u> – if you are discharged from the hospital before these visits, you may be asked to return to clinic if it is safe to do so.

- Your vital signs will be recorded.
- You will also have blood drawn for routine laboratory testing. About 3 tablespoons of blood will be collected.
- A nasal or oral swab will be taken for testing of the virus again. This procedure will be done for research purposes only. The specimen will be stored for future use. An appendix at the end of this form discusses what may happen to your specimen.

<u>Day 30/End of Study</u> – if you are discharged from the hospital before this visit, you may be asked to return to clinic if it is safe to do so.

- Your vital signs will be recorded.
- Blood will be drawn for routine laboratory testing. About 3 tablespoons of blood will be collected.

## 6. Benefits to Subjects:

If the medications work, you may see improvement in the symptoms of COVID-19 infection and have a shorter recovery time. However, you may not receive a health benefit by participating in

 LSUHSC-NO IRB#: 20-047

Consent Rev. date: 03Apr2020 Protocol Revision #: 31Mar2020, v10

this study. The information we collect during this study may help us to treat COVID-19 infection or other viral infections in the future.

## 7. Risks to Subject:

As with all medications and procedures, there are some known side effects that may occur during your treatment.

# **Hydroxychloroquine**

## Common Side Effects:

- nausea
- vomiting
- stomach/abdominal pain or cramps
- loss of appetite
- weight loss
- diarrhea
- dizziness
- spinning sensation

- headache
- ringing in your ears
- mood changes
- nervousness
- irritability
- skin rash
- itching
- hair loss

#### Less Common/Rare Side Effects:

\_

- abnormal electrocardiogram (ECG): a condition called prolonged QT can occur and may lead to heart arrhthymias (abnormal heartbeat)
- side effects affecting vision: blurred vision, light sensitivity, seeing halos around lights, and retinopathy which may occur in 4% of patients with long-term use
- side effects affecting nervous system: twitching, uncontrolled movement, loss of balance or coordination, confusion, unusual thoughts or behavior, and seizures (convulsions)
- Other less common side effects include:
  - Muscle weakness
  - Pale skin

- Easy bruising
- o Bleeding

## Azithromycin

#### Common Side Effects:

- diarrhea or loose stools
- nausea

## Less Common/Rare Side Effects:

- stomach upset
- vomiting
- constipation
- dizziness
- tiredness
- headache

- stomach/abdominal pain
- vaginal itching or discharge
- nervousness
- sleep problems (insomnia)
- skin rash or itching
- ringing in the ears
- hearing problems

 LSUHSC-NO IRB#: 20-047

Consent Rev. date: 03Apr2020 Protocol Revision #: 31Mar2020, v10

- or decreased sense of taste or smell
- abnormal electrocardiogram (ECG): a condition called prolonged QT can occur and may lead to heart arrhthymias (abnormal heartbeat)

<u>Blood draws</u> – you may experience pain from the needle puncture, bruising, bleeding, fainting, or rarely, infection from having blood drawn. Every effort will be made to minimize discomfort.

<u>Electrocardiogram (ECG)</u> – you may experience skin irritation from the gel or electrode pads used during an ECG.

<u>Chest X-ray</u> – the amount of radiation from a chest X-ray is not more than you would experience in everyday life.

There is a risk that someone could trace the information in a central database back to you. Even without your name or other identifiers, your genetic information is unique to you. The researchers believe the chance that someone will identify you is very small, but the risk may change in the future as people come up with new ways of tracing information.

## 8. Alternatives to Participation in the Study:

The alternative is not to participate.

## 9. Subject Removal:

The researcher may stop you from taking part in this study if at any time it is believed to be in your best interest; if you do not follow the study procedures; if the study is stopped. You could be taken off the study if your health worsens; if another treatment option appears to be appropriate; or for any other cause which prevents your continuing in the study.

## 10. Subject's Right to Refuse to Participate or Withdraw:

Participation is voluntary. Refusal to participate will involve no penalty or loss of benefits to which you are otherwise entitled, and you may discontinue participation at any time without penalty or loss of benefits to which you are otherwise entitled. You may refuse to participate or withdraw from the study at any time without jeopardizing, in any way, your medical treatment at this institution in the present or future. Information already collected about you and sent to the sponsor will still be used. Tell the researcher if you are thinking about withdrawing from the study so that you may do so safely. If you decide not to continue participation in the study you should seek medical advice for alternatives. Should significant new findings take place during the course of the research that may relate to your willingness to continue participation, that information will be provided to you.

# 11. Subject's Right to Privacy:

If the results of the study are published the privacy of subjects will be protected and they will not be identified in any way. Your personal information may be disclosed if required by law.

A Federal law, called the Genetic Information Nondiscrimination Act (GINA), generally makes it illegal for health insurance companies, group health plans, and most employers to discriminate

 LSUHSC-NO IRB#: 20-047

Consent Rev. date: 03Apr2020 Protocol Revision #: 31Mar2020, v10

against you based on your genetic information. This law generally will protect you in the following ways:

- Health insurance companies and group health plans may not request your genetic information that we get from this research.
- Health insurance companies and group health plans may not use your genetic information that we get from this research when making decisions regarding your eligibility or premiums.
- Employers with 15 or more employees may not use your genetic information that we get from this research when making a decision to hire, promote, or fire you or when setting the terms of your employment.

Louisiana law prohibits discrimination in employment or insurability based on your genetic information. Your genetic information is considered your property and no insurer or employer may obtain genetic information or a DNA sample without first obtaining your written consent. (LA Statute RS22:1023 and RS23:368).

#### 12. Release of Information:

Organizations that may inspect and/or copy your study-related medical records for quality assurance and data analysis include: the LSUHSC-NO Institutional Review Board, the UMC Office of Research, the doctors listed on page 1 of this consent form and their staff, and the Food and Drug Administration (FDA). While every effort will be made to maintain your privacy, absolute confidentiality cannot be guaranteed. Records will be kept private to the extent allowed by law.

#### 13. Financial Information:

Participation in this study will not result in any extra charges above and beyond those routinely incurred by patients with similar conditions. The study drugs will be provided by UMCNO. Any expenses not paid by insurance will be billed to you.

The principal investigator will arrange for medical care for any emergency medical problem that you may experience as a direct result of your participation in this research. This will be provided on a fee-for-service basis. There are not funds available to pay for any disability that results or for damages such as lost wages, etc.

You will not be paid for your participation as reimbursement for your time and travel.

If commercial products or other valuable discoveries result from this research project, these products and discoveries could be patented, licensed, or otherwise developed for commercial sale by UMCNO, the investigators, or their designees. If this should occur, we will not provide financial compensation to you, or share with you the patent rights, other ownership right, or rights to control any resulting commercial products and discoveries that my result from this research project.

## 14. Signatures:

The study has been discussed with me and all my questions have been answered. Additional

 LSUHSC-NO IRB#: 20-047

Consent Rev. date: 03Apr2020 Protocol Revision #: 31Mar2020, v10

questions regarding the study should be directed to the investigators listed on page 1 of this consent form. If I have questions about subject's rights, or want to discuss problems, concerns or questions, or obtain information or offer input, I can contact the Chancellor of the LSU Health Sciences Center New Orleans at (504) 568-4801. I agree with the terms above, acknowledge I have been given a copy of the consent form, and agree to participate in this study. I have not waived any of my legal rights by signing this consent form.

| Printed name of Subject | · |
|---|---|
| Signature of Subject or LAR | Date |
| Printed Name of LAR (if subject is unable to s | sign) |
| Consent Administered by | Date |
| Printed Name | |
| Printed Name of Witness to consent (if consen | nt administered remotely) |
| Signature of Witness to consent (if consent add | <br>ministered remotely) |
| | e subject is unable to read. I certify that I have read ed that by completing the signature line above the |
| Signature of Reader | Date |
| Printed Name | |

 LSUHSC-NO IRB#: 20-047 Consent Rev. date: 03Apr2020 Protocol Revision #: 31Mar2020, v10

| Signature of Witness | Date |
|----------------------|------|
| Printed Name | |

 LSUHSC-NO IRB#: 20-047

Consent Rev. date: 03Apr2020 Protocol Revision #: 31Mar2020, v10

## Appendix: Biospecimens stored for future unspecified use

Donating your tissue and/or blood (called bio-specimens) for future, unspecified research is an important decision. Your bio-specimens may be used for research concerning your condition or for other unrelated diseases. This important research may help future patients with their health problems. However, you should consider not only this potential benefit but other important information before agreeing to donate tissue and/or blood.

For example, you should be aware of the following:

- 1. Tissue and/or blood samples will be stored and used for an unknown period of time.
- 2. General, identifiable health information may be included with your bio-specimens. In this case, a link will exist between your health information and the donated tissue and/or blood and the donation would not be considered de-identified (or anonymous).
- 3. This information and tissue samples may be shared with a wide range of researchers and institutions.
- 4. Your tissue samples may be used for research other than cancer research.
- 5. Your tissue may be used for genetic analyses allowing your identity to be known.
- 6. There is the possibility of your samples and information being used for the development of commercially available treatments or tests.
- 7. Future research may use techniques not currently available or understood.
- 8. Now and/or in the future, certain kinds of sensitive or controversial research may be conducted with your bio-specimens. For example certain types of reproductive research may be conducted such as cloning or the development of human stem cells.

The material above has been presented to and discussed with the potential subject.

| I have read | I the conditions above and agree to allow storage of my biospecimens for future use. |
|---|---|
| <br>Initial | _ □ YES |
| <br>Initial | _□ NO |